CLINICAL TRIAL: NCT04175899
Title: Effectiveness of Pharmacist Intervention on Capecitabine Relative Dose Intensity, Adherence, Knowledge & Safety Among Cancer Patients in Malaysia.
Acronym: POCCP1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Malaysia (Other Government)
Collaborators: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Tajunisah Mohamed Eusoff, Principle Investigator, Ministry of Health, Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: POCCP1 v1.3_10July19; NMRR-18-3634-44321 (IIR) (Other: Medical Research & Ethics Committee, Malaysia)
Record Dates: First submitted 2019-11-19; First posted 2019-11-25 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor, Adult
Keywords: Capecitabine; Pharmacist Intervention; Adherence; Relative Dose Intensity; Medication Knowledge; Safety
MeSH Terms: interventions — Pharmaceutical Services

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- POCCP (Pharmacist-led Oral Chemo Care Program) (Experimental): Intervention Group :
  Subjects undergo structured intensified pharmaceutical care program (POCCP) led by oncology experienced pharmacist (run alongside oncologist patient review at the clinic or daycare) in addition to Current Standard Best Care (SBC)
  Interventions: Other: Pharmacist-led Oral Chemo Care Program (POCCP)
- SBC (Current Standard Best Care) (No Intervention): Control Group :
  Subjects undergo usual procedure which is Current Standard Best Care (SBC) for oral chemotherapy treatment which includes pre-chemotherapy review by doctor and prescribing of chemotherapy and supportive medications according to patient's chemotherapy protocol at each visit. Subsequently the patients will collect their prescribed oral medications at the ambulatory pharmacy counter according to the standard procedure of medication dispensing which includes prescription screening, medication filling, double checking, dispensing and counselling at the pharmacy counter as per usual practice of pharmaceutical care of patients.

INTERVENTIONS:
Other: Pharmacist-led Oral Chemo Care Program (POCCP) — Structured intensified pharmaceutical care program for patients ongoing oral chemotherapy treatment.
  Led by oncology experienced clinical pharmacist and run alongside oncologist patient review at the clinic or daycare.
  It utilizes structured educational material (for patients) and monitoring guideline or checklists (for pharmacists) during provision of service at each clinic visit such as patient education, pre-treatment review, medication reconciliation, prescription screening (dose, regime, supportive meds), adherence, adverse drug event monitoring and treatment recommendations on basis of agreed protocols.
  Pharmacist scheduled additional review within 1-week interval of start of oral chemotherapy at clinic or via phone call (according to patient's preference) will also be conducted to review patients taking their oral medications at home, assess adherence and symptom experienced to provide individualized recommendations or support to patients.
  Other Names: Pharmaceutical Care
  Arms: POCCP (Pharmacist-led Oral Chemo Care Program)

SUMMARY:
Over the past decade, oral administration of chemotherapy has significantly increased and is anticipated to continue to grow. Despite the conveniences, these oral regimens can be complex and pose challenge to patient adherence. Further safety concerns are warranted due to insufficient patient education, general perception of reduced toxicity with oral treatment, improper prescribing practice, and the lack of monitoring of observable adverse effects.

Therefore, effective medication counselling and patient education is vital to empower patients and their caregivers to increase adherence and safely managed medication to achieve optimal treatment outcome.

This study aims to evaluate the effectiveness of pharmacist intervention with structured oral chemotherapy education and patient monitoring on capecitabine treatment effectiveness (Relative Dose Intensity (RDI), Adherence and Persistence), safety outcomes (Adverse Event, Drug Related Problem and Health service utilization) and chemotherapy knowledge and self-efficiency among cancer patient care in Penang, a northern state oncology referral centre.

There are numerous published studies of pharmaceutical care implementations focusing mainly on in-patient setting and currently evolving in ambulatory cancer patients especially in western countries compared to Asian region. However systematic reviews show major gap still exist with paucity of scientific evidence on the effectiveness of therapeutic educational interventions for improving patient safety and adherence to oral chemotherapy mainly due to study design and method that are unable to strongly prove the outcome.

Hence highlighting the novelty and significance for this research using randomized controlled design, standardized & validated tools for multimodal pharmacist intervention, long-term clinical outcome such as RDI with longitudinal assessment till treatment completion.

ELIGIBILITY:
Inclusion Criteria:

Patients will be screened according to the inclusion criteria below;

1. Adult patients (≥ 18 years old)
2. Ambulatory patients (daycare or out-patient oncology department clinic)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 2 or below,
4. Diagnosis of Colorectal, Breast, Stomach cancer
5. Newly started on oral Capecitabine (Xeloda) either as a single agent or in combination with other intravenous chemotherapy
6. Adjuvant or metastatic treatment intent
7. Patients who have given written consent to participate in the study.

Exclusion Criteria:

The following patients will be excluded from the study:

1. Patients who are ongoing in other clinical trial,
2. Patients with dementia, cognitive disability, mental retardation, Alzheimer's or Parkinson's
3. Patients on concurrent radiotherapy regime with capecitabine.
4. Patients who are unable to respond to questions or could not speak and understand Malay, English or Chinese language
5. Patients who are unable to complete the questionnaires with minimal assistance from researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Relative Dose Intensity - End of Treatment | 6 months
  RDI will be assessed at the end of Cycle 8 (each cycle is 21 days). Relative dose intensity (RDI), defined as the total dose administered divided by the total dose specified by the corresponding standard regimen.
Relative Dose Intensity - Mid Treatment | 3 months
  RDI will be assessed at the end of Cycle 4 (each cycle is 21 days). Relative dose intensity (RDI), defined as the total dose administered divided by the total dose specified by the corresponding standard regimen.
Daily Adherence | 6 months
  Daily Adherence will be assessed at the end of Cycle 8 (each cycle is 21 days). The daily adherence level determined by the pill count, patient diary record at each visit, which considered both the correct administration of capecitabine twice daily for 14 days and correct non-administration of any dose on rest days to be determined as adherent throughout the 21 day cycle.

SECONDARY OUTCOMES:
Persistence to Treatment | 6 months
  Persistence to Treatment defined as percentage of patient completed 8 cycle of treatment (each cycle is 21 days).
Medication Adherence Report Scale (MARS-5) C1 | 3 weeks
  MARS-5 score will be assessed at the end of Cycle 1 (each cycle is 21 days). Medication Adherence Report Scale (MARS-5) Questionnaire consists of five questions on patterns of nonadherent behaviour to assess patients self-reported adherence to oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 25 whereby a higher scores means better adherence.
Medication Adherence Report Scale (MARS-5) C4 | 3 months
  MARS-5 score will be assessed at the end of Cycle 4 (each cycle is 21 days). Medication Adherence Report Scale (MARS-5) Questionnaire consists of five questions on patterns of nonadherent behaviour to assess patients self-reported adherence to oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 25 whereby a higher scores means better adherence.
Medication Adherence Report Scale (MARS-5) C8 | 6 months
  MARS-5 score will be assessed at the end of Cycle 4 (each cycle is 21 days). Medication Adherence Report Scale (MARS-5) Questionnaire consists of five questions on patterns of nonadherent behaviour to assess patients self-reported adherence to oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 25 whereby a higher scores means better adherence.
Capecitabine Medication Taking Behavior Questionnaire C1 | 3 weeks
  Capecitabine Medication Taking Behavior (CMTB) will be assessed at the end of Cycle 1 (each cycle is 21 days).
  The questionnaire consists of four questions to further identify aspects of patients non-adherence, their medication-taking and medication-stopping behavior specific for oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 20 whereby a higher scores means better adherence.
Capecitabine Medication Taking Behavior Questionnaire C4 | 3 months
  Capecitabine Medication Taking Behavior (CMTB) will be assessed at the end of Cycle 4 (each cycle is 21 days).
  The questionnaire consists of four questions to further identify aspects of patients non-adherence, their medication-taking and medication-stopping behavior specific for oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 20 whereby a higher scores means better adherence.
Capecitabine Medication Taking Behavior Questionnaire C8 | 6 months
  Capecitabine Medication Taking Behavior (CMTB) will be assessed at the end of Cycle 8 (each cycle is 21 days).
  The questionnaire consists of four questions to further identify aspects of patients non-adherence, their medication-taking and medication-stopping behavior specific for oral capecitabine. Scoring is on a 5-point Likert scale and total score range between 5 and 20 whereby a higher scores means better adherence.
Change in Chemotherapy Knowledge & Self-Efficiency C1 | 3 weeks
  Change in Chemotherapy Knowledge & Self-Efficiency will be assessed at the end of Cycle 1 (3 weeks) from baseline (week 0). Each cycle is 21 days Patients chemotherapy knowledge and self-efficiency level will be assessed using a structured question set.
Change in Chemotherapy Knowledge & Self-Efficiency C4 | 3 months
  Change in Chemotherapy Knowledge & Self-Efficiency will be assessed at the end of Cycle 4 (3 months) from baseline (week 0). Each cycle is 21 days Patients chemotherapy knowledge and self-efficiency level will be assessed using a structured question set.
Change in Chemotherapy Knowledge & Self-Efficiency C8 | 6 months
  Change in Chemotherapy Knowledge & Self-Efficiency will be assessed at the end of Cycle 8 (6 months) from baseline (week 0). Each cycle is 21 days Patients chemotherapy knowledge and self-efficiency level will be assessed using a structured question set.
Change in Adverse Drug Events (ADE) - Toxicity Score | 6 months
  Change in Toxicity Score will be assessed at the end of Cycle 8 (6 months) from baseline (week 0). Each cycle is 21 days Incidence and severity grading of adverse events related to chemotherapy, will be measured by the reviewing doctor for the duration of treatment follow-up using a standardized ADE monitoring checklist based on the National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) v4.0 grading scale.
Drug Related Problem (DRP) and Pharmacist Intervention | 6 month
  Frequency of DRPs identified during the study will be reported using the Pharmaceutical Care Network Europe (PCNE) classification scheme v8.01
Health service utilization | 6 month
  Frequency of hospital services utilizations of the patients will be measured for emergency department visit, unplanned oncology clinic or outpatient visits, hospital admissions or had phone calls to oncology clinic.

CONTACTS AND LOCATIONS:
Overall Officials: Balamurugan Tangiisuran, PhD, Study Director — Universiti Sains Malaysia
Locations (1):
- Hospital Pulau Pinang, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No